CLINICAL TRIAL: NCT01333527
Title: Early Mobilization Following Arthroscopic Rotator Cuff Repair: a Randomized Controlled Trial
Brief Title: Early Mobilization Following Arthroscopic Rotator Cuff Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RES0005824
Record Dates: First submitted 2011-04-08; First posted 2011-04-12 (Estimated); Results first posted 2021-09-13 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Rotator Cuff Tear
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Suburethral Slings

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (early ROM) (Experimental): Group A (early ROM) will use the sling for comfort only
  Interventions: Procedure: No Sling
- Group B (usual care) (Active Comparator): Group B (usual care) will be immobilized in a sling for 6 weeks.
  Interventions: Procedure: Sling

INTERVENTIONS:
Procedure: No Sling — Early range of motion
  Arms: Group A (early ROM)
Procedure: Sling — Patients will use the sling for 6 weeks, as per usual care
  Arms: Group B (usual care)

SUMMARY:
Shoulder rotator cuff (RC) tears are a significant cause of pain and disability. Surgery is done to reconnect the torn RC tendon(s) to the bone. The goals of RC surgery are to decrease pain, and to increase range of motion (ROM) and strength. This is done arthroscopically; through a small incision in the patient's shoulder. After surgery, patients are usually placed in a sling for up to 6 weeks to protect the repaired shoulder tendons. During this time, ROM exercises are only done by using the un-operated arm for assistance. Voluntary or active shoulder movement is usually not permitted to allow the repaired tendons to heal. Unfortunately, some patients develop shoulder stiffness while wearing the sling, which can delay rehabilitation. Any delays in rehabilitation may result in reduced shoulder function, a slower return-to-work or daily activities, and may also impact the health care system, through increased use and cost of rehabilitation.

This study's purpose is to determine if patients can safely stop wearing their sling as early as pain and comfort allow following RC surgery. A total of 200 patients (100 per group) will be randomly assigned to one of two study groups:

Patients in Group A (accelerated rehab) will wear their sling for comfort only following surgery. Self-assisted ROM exercises are allowed at any time. This means that patients may stop wearing their sling if pain and comfort allow, and start active movement for activities of daily living only.

Patients in Group B (standard rehab) will wear their sling for 6 weeks. Like in group A, self-assisted ROM exercises are allowed at any time, but active movement will not be allowed until 6 weeks after surgery. Patients in both groups will be given the same self-assisted ROM exercises after surgery.

Patients who agree to participate in the study will see their surgeon and the study physical therapist/research coordinator on 6 occasions (pre-surgery, 2 weeks, 6 weeks, 3, 6, 12 months post-surgery). Each visit will take about 30 minutes and will include a ROM assessment, strength assessment (as appropriate) and disease-specific quality of life questionnaires. Patients will also undergo an Ultrasound exam to verify that their RC repair is intact at 12-months. Differences in ROM, strength, questionnaire scores, RC integrity, and adverse events will be examined between the two groups. Differences will also be examined according to RC tear size and patient characteristics.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is over 18 years of age
2. Patient has attempted non-operative treatment (i.e. physical therapy consisting of progressive ROM, strengthening, and postural exercises)
3. Patient has a full-thickness tear of the supraspinatus and/or infraspinatus, as confirmed by appropriate diagnostic imaging (MRI, Arthrogram, Ultrasound)

Exclusion Criteria:

1. Patient has a full-thickness tear of the subscapularis and/or teres minor
2. Patient has undergone previous RC surgery to the affected shoulder
3. Patient has major joint trauma, infection, or avascular necrosis
4. Patient has chronic dislocation, inflammation, or degenerative glenohumeral arthropathy
5. Patient has evidence of significant cuff arthropathy (superior glenohumeral translation and/or acromial erosion, as diagnosed by diagnostic imaging)
6. Patient has a psychiatric illness, cognitive impairment, or other health condition (i.e. visual impairment) which precludes informed consent or renders the patient unable to complete study questionnaires
7. Patient has a major medical illness where life expectancy is less than 2 years
8. Patient does not speak/read/understand English
9. Patient has no fixed address or means of contact
10. Surgeon or patient has decided to cancel surgery
11. Surgeon concludes that an arthroscopic repair is not appropriate at time of surgery (based on RC tear characteristics or concomitant shoulder pathology)
12. Patient unwilling to complete necessary follow-ups

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2011-04; Primary Completion 2015-04 (Actual); Study Completion 2018-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Sheps, MD,MSc,FRCSC, Principal Investigator — University of Alberta
Locations (1):
- Glen Sather Sports Medicine clinic, Edmonton, Alberta, Canada

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Withdrew following randomization (n=5)
  Reasons:
  n=4 : Had Abduction pillow n=1: Excluded at surgery
Period: Overall Study
Arm/Group | Group A (Early ROM) | Group B (Usual Care)
Started | 105 | 106
Completed | 87 | 89
Not Completed | 18 | 17

BASELINE CHARACTERISTICS:
Groups:
- Group A (Early ROM): Group A (early ROM) used the sling for comfort only
- Group B (Usual Care): Group B (usual care) used the sling for 6 weeks
- Total: Total of all reporting groups
Arm/Group | Group A (Early ROM) | Group B (Usual Care) | Total
Number analyzed (Participants) | 103 | 103 | 206
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (8.3) | 56.2 (10.1) | 55.85 (9.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 37 | 75
  Male | 65 | 66 | 131
Region of Enrollment [Number; unit: participants]
  Canada | 103 | 103 | 206
Range of Motion [Mean (Standard Deviation); unit: degrees] — Measured flexion, abduction, external rotation in 90 degrees abduction [ER(90)], internal rotation in 90 degrees abduction [IR(90)], horizontal adduction, scaption, degrees with a goniometer by the same tester throughout
  degrees
    Flexion_Baseline | 132.1 (30.7) | 127.7 (35.6) | 129.91 (33.21)
    Abduction_Baseline | 122 (36.6) | 118.9 (39.8) | 120.44 (38.18)
    External rotation 90 degrees abduction | 61.0 (34.8) | 61.6 (31.8) | 61.3 (33.23)
    Internal rotation with 90 degrees abduction | 30.8 (19.1) | 33.3 (17.8) | 32.08 (18.43)
Western Ontario Rotator Cuff Index (WORC) [Mean (Standard Deviation); unit: percentage] — a 5-part (physical symptoms, sports/recreation, work, lifestyle, emotions) 21-item disease specific questionnaire. Measured in percentage. 0% = worst, 100 % = best
  percentage | 38.9 (18.5) | 40.6 (17.2) | 39.75 (17.88)
Pain scale (Visual Analogue) [Mean (Standard Deviation); unit: units on a scale] — Shoulder pain at rest, with activity and at night were measured using a visual analogue scale of 0-10 (no pain to severe pain)
  units on a scale
    pain at rest | 3.1 (2.3) | 2.9 (2.4) | 3.0 (2.34)
    pain with activity | 6.1 (2.4) | 5.7 (2.4) | 5.88 (2.39)
    pain at night | 4.8 (2.6) | 4.3 (2.7) | 4.57 (2.68)
Strength (dynamometer microFIT3) [Mean (Standard Deviation); unit: pounds] — strength was measured in pounds of force using a dynamometer (microFET3, Hoggan Health Industries, West Jordan, UT). Isometric shoulder flexion, abduction, were measured with the arm in neutral abduction and elbow at 90 degrees flexion. External and internal rotation were measured in 90 degrees of abduction. Peak values were recorded during each contraction which was held for 3 seconds. Values were expressed as raw values as well as proportional to the unaffected shoulder.
  pounds
    flexion | 19.2 (10.9) | 20.1 (12.3) | 19.66 (11.6)
    abduction | 18.0 (9.8) | 18.0 (9.8) | 18.0 (9.7)
    External rotation in abduction | 11.2 (8.3) | 11.9 (9.3) | 11.54 (8.8)
    internal rotation in abduction | 17.6 (12.3) | 19.4 (14.0) | 18.53 (13.21)
    horizontal adduction | 17.4 (11.8) | 20.2 (13.3) | 18.8 (12.6)
    scaption | 13.99 (6.92) | 14.14 (7.55) | 14.07 (7.23)
Short-Form 36-Item Health Survey (SF-36) [Mean (Standard Deviation); unit: units on a scale] — Quality of life questionnaire that looks at physical functioning, Role-physical, bodily pain, general health, vitality, social function, role-emotional, mental health on a scale of worst to best. It is scored between 0 (no disability) and 100(very disable).
  units on a scale
    physical functioning | 72.1 (15.8) | 71.7 (16.3) | 71.87 (16.02)
    role physical | 33.5 (39.2) | 35.7 (36.8) | 34.59 (37.96)
    Bodily pain | 44.7 (17.2) | 46.7 (18.9) | 45.67 (18.03)
    general health | 78.8 (15.8) | 76.0 (17.6) | 77.39 (16.74)
    vitality | 61.0 (20.7) | 62.2 (18.1) | 61.62 (19.4)
    social function | 79.6 (21.9) | 76.1 (22.1) | 77.85 (22.02)
    role emotional | 78.6 (37.3) | 80.3 (33.8) | 79.45 (35.51)
    mental health | 78.4 (15.1) | 77.7 (13.7) | 78.08 (14.41)
Surgical Characteristics [Mean (Standard Deviation); unit: cm]
  Mean length of tear Anteroposterior | 2.1 (1.1) | 2.1 (1.0) | 2.1 (1.04)
  Mean length of tear Mediolateral | 1.9 (1.1) | 1.9 (1.1) | 1.9 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Western Ontario Rotator Cuff Index (WORC)
Description: a 5-part (physical symptoms, sports/recreation, work, lifestyle, emotions) 21-item disease specific questionnaire. Measured in percentage. 0% = worst, 100 % = best
Time Frame: Baseline, 6 weeks, 3 months, 6 months, 12 months and 24 months
Measure: Mean (Standard Deviation); unit: percentage
Groups:
- Group A (Early ROM): Group A (early ROM) will use the sling for comfort only
  No Sling: Early range of motion
  Overall number of Baseline participants: 103. >18 years, continuous Sex: male and female Region of enrollment
- Group B (Usual Care): Group B (usual care) will be immobilized in a sling for 6 weeks.
  Sling: Patients will use the sling for 6 weeks, as per usual care
  Overall number of Baseline participants 103 >18 years, continuous Sex: male and female Region of enrollment
Arm/Group | Group A (Early ROM) | Group B (Usual Care)
Number analyzed (Participants) | 87 | 89
percentage
  Baseline | 39.2 (18.4) | 40.2 (17.3)
  6 weeks | 44.5 (16.6) | 40.7 (14.0)
  3 months | 61.4 (19.0) | 63.7 (17.6)
  6 months | 78.6 (16.8) | 79.6 (15.2)
  12 months | 87.6 (14.1) | 88.6 (13.1)
  24 months | 89.4 (13.4) | 89.8 (13.4)

2. Primary Outcome: Range of Motion (ROM)
Description: Measured flexion, abduction, external rotation in 90 degrees abduction [ER(90)], internal rotation in 90 degrees abduction [IR(90)], horizontal adduction, scaption, degrees with a goniometer by the same tester throughout
Time Frame: baseline, 6 weeks, 3 months, 6 months, 12 months and 24 months
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Group A (Early ROM) | Group B (Usual Care)
Number analyzed (Participants) | 87 | 89
degrees
  Forward Flexion baseline | 131.5 (30.0) | 127.4 (34.9)
  Forward Flexion 6 weeks | 90.0 (33.4) | 78.9 (34.5)
  Forward Flexion 3 months | 125.5 (28.5) | 121.0 (30.1)
  Forward Flexion 6 months | 142.3 (22.6) | 141.3 (22.6)
  Forward Flexion12 months | 150.9 (12.6) | 149.0 (19.9)
  Forward Flexion 24 months | 155.5 (12.7) | 152.2 (18.5)
  Abduction baseline | 121.1 (36.0) | 118.6 (39.4)
  Abduction 6 weeks | 75.4 (36.8) | 67.1 (32.9)
  Abduction 3 months | 119.1 (31.3) | 116.0 (37.6)
  Abduction 6 months | 139.4 (23.5) | 139.5 (27.6)
  Abduction 12 months | 150.0 (15.3) | 148.4 (22.4)
  Abduction 24 months | 153.5 (14.6) | 152.2 (21.9)
  External Rotation in Abduction Baseline | 62.2 (34.1) | 61.6 (31.6)
  External Rotation in Abduction 6 weeks | 22.0 (29.2) | 19.5 (28.8)
  External Rotation in Abduction 3 months | 53.0 (27.6) | 44.2 (28.8)
  External Rotation in Abduction 6 months | 67.6 (21.0) | 62.9 (21.6)
  External Rotation in Abduction 12 months | 75.3 (16.2) | 70.6 (18.8)
  External Rotation in Abduction 24 months | 76.0 (14.8) | 71.5 (17.8)
  Internal rotation in abduction baseline | 30.6 (18.6) | 33.2 (17.6)
  Internal rotation in abduction 6 weeks | 14.1 (18.6) | 11.8 (16.6)
  Internal rotation in abduction 3 months | 30.2 (15.2) | 25.9 (16.3)
  Internal rotation in abduction 6 months | 35.9 (12.1) | 35.5 (12.2)
  Internal rotation in abduction 12 months | 39.0 (12.4) | 40.1 (14.4)
  Internal rotation in abduction 24 months | 40.9 (12.0) | 38.7 (12.4)
  Horizontal adduction baseline | 13.2 (9.2) | 14.4 (10.3)
  Horizontal adduction 6 weeks | 8.2 (10.0) | 6.4 (9.3)
  Horizontal adduction 3 months | 14.9 (9.7) | 13.0 (9.7)
  Horizontal adduction 6 months | 19.4 (13.5) | 18.1 (9.9)
  Horizontal adduction 12 months | 19.1 (10.4) | 18.9 (10.4)
  Horizontal adduction 24 months | 20.4 (10.5) | 19.5 (11.5)
  Scaption baseline | 124.6 (31.3) | 123.6 (34.8)
  Scaption 6 weeks | 80.4 (33.1) | 75.8 (36.3)
  Scaption 3 months | 120.7 (28.0) | 118.5 (31.0)
  Scaption 6 months | 138.0 (21.4) | 137.9 (23.6)
  Scaption 12 months | 148.7 (11.7) | 146.7 (20.2)
  Scaption 24 months | 151.7 (12.8) | 149.7 (18.8)

3. Secondary Outcome: Strength
Description: strength was measured in pounds of force using a dynamometer (microFET3, Hoggan Health Industries, West Jordan, UT). Isometric shoulder flexion, abduction, were measured with the arm in neutral abduction and elbow at 90 degrees flexion. External and internal rotation were measured in 90 degrees of abduction. Peak values were recorded during each contraction which was held for 3 seconds. Values were expressed as raw values.
Time Frame: Baseline, 6 months, 12 months, 24 months
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Group A (Early ROM) | Group B (Usual Care)
Number analyzed (Participants) | 87 | 89
pounds
  Flexion baseline | 19.6 (10.9) | 19.8 (12.3)
  Flexion 6 months | 26.3 (12.6) | 27.1 (10.8)
  Flexion 12 months | 29.7 (13.7) | 31.0 (12.7)
  Flexion 24 months | 28.3 (11.5) | 29.1 (11.7)
  Abduction baseline | 18.6 (10.0) | 17.8 (10.1)
  Abduction 6 months | 23.2 (10.1) | 23.2 (9.3)
  Abduction 12 months | 26.8 (10.7) | 26.9 (10.5)
  Abduction 24 months | 26.9 (9.6) | 28.2 (10.6)
  External rotation in abduction baseline | 11.5 (8.4) | 11.9 (9.6)
  External rotation in abduction 6 months | 18.2 (9.4) | 18.7 (10.1)
  External rotation in abduction 12 months | 23.3 (12.5) | 24.0 (12.3)
  External rotation in abduction 24 months | 25.1 (12.5) | 24.8 (11.8)
  Internal rotation in abduction baseline | 18.1 (12.7) | 19.5 (14.1)
  Internal rotation in abduction 6 months | 27.1 (14.5) | 26.7 (12.5)
  Internal rotation in abduction 12 months | 30.9 (15.2) | 32.3 (14.4)
  Internal rotation in abduction 24 months | 30.6 (13.1) | 31.3 (13.4)
  Horizontal Adduction baseline | 17.7 (12.2) | 20.0 (13.4)
  Horizontal Adduction 6 months | 25.7 (12.1) | 25.4 (10.7)
  Horizontal Adduction 12 months | 28.1 (11.3) | 28.4 (11.6)
  Horizontal Adduction 24 months | 27.9 (9.8) | 28.2 (11.1)
  Scaption baseline | 14.2 (7.1) | 13.9 (7.2)
  Scaption 6 months | 16.4 (6.9) | 16.3 (6.5)
  Scaption 12 months | 19.8 (7.3) | 19.1 (7.0)
  Scaption 24 months | 20.6 (7.0) | 19.7 (7.2)

4. Secondary Outcome: The Short Form (36) Health Survey
Description: The Short Form (36) Health Survey is a quality of life questionnaire that looks at eight scales: physical functioning, Role-physical, bodily pain, general health, vitality, social function, role-emotional, mental health. Each scale ranges between 0 (completely disable) to 100 (completely able).
Time Frame: baseline, 6 weeks, 3 months, 6 months, 12 months and 24 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A (Early ROM) | Group B (Usual Care)
Number analyzed (Participants) | 87 | 89
units on a scale
  physical functioning baseline | 72.8 (15.2) | 71.3 (16.7)
  physical functioning 6 weeks | 68.2 (14.2) | 64.7 (15.2)
  physical functioning 3 months | 75.0 (15.9) | 73.7 (16.3)
  physical functioning 6 months | 84.4 (14.1) | 82.7 (18.1)
  physical functioning 12 months | 89.3 (13.2) | 86.3 (18.2)
  physical functioning 24 months | 86.8 (15.4) | 85.7 (16.9)
  role physical baseline | 33.2 (39.1) | 36.6 (37.7)
  role physical 6 weeks | 14.7 (28.8) | 10.6 (25.4)
  role physical 3 months | 40.9 (42.7) | 37.5 (41.2)
  role physical 6 months | 71.1 (37.6) | 65.6 (40.2)
  role physical 12 months | 86.1 (29.6) | 79.8 (35.8)
  role physical 24 months | 81.8 (33.6) | 74.4 (38.8)
  bodily pain baseline | 43.5 (16.4) | 46.3 (18.6)
  bodily pain 6 weeks | 50.2 (22.8) | 45.5 (24.0)
  bodily pain 3 months | 62.5 (22.5) | 66.5 (20.5)
  bodily pain 6 months | 69.5 (17.8) | 71.7 (19.2)
  bodily pain 12 months | 74.6 (20.0) | 75.5 (20.8)
  bodily pain 24 months | 73.2 (22.2) | 76.7 (22.7)
  General Health baseline | 79.0 (15.4) | 76.0 (17.9)
  General Health 6 weeks | 78.0 (17.1) | 77.7 (17.0)
  General Health 3 months | 77.6 (14.7) | 79.3 (17.0)
  General Health 6 months | 81.1 (13.5) | 79.7 (15.4)
  General Health 12 months | 80.3 (14.6) | 80.1 (15.7)
  General Health 24 months | 78.8 (17.3) | 77.2 (20.0)
  Vitality baseline | 61.0 (20.3) | 63.2 (18.2)
  Vitality 6 weeks | 58.9 (18.8) | 57.3 (19.2)
  Vitality 3 months | 65.9 (18.1) | 68.0 (16.7)
  Vitality 6 months | 70.4 (15.4) | 72.9 (14.0)
  Vitality 12 months | 73.2 (15.4) | 73.9 (14.0)
  Vitality 24 months | 70.7 (19.9) | 73.9 (16.3)
  Social function baseline | 79.0 (22.2) | 76.5 (22.1)
  Social function 6 weeks | 70.0 (26.3) | 61.7 (26.1)
  Social function 3 months | 82.4 (20.0) | 81.1 (20.6)
  Social function 6 months | 90.5 (16.5) | 90.4 (15.4)
  Social function 12 months | 90.4 (17.1) | 91.1 (17.2)
  Social function 24 months | 86.4 (21.3) | 88.7 (18.8)
  role emotional baseline | 80.2 (36.2) | 81.4 (33.9)
  role emotional 6 weeks | 65.9 (42.7) | 64.2 (43.0)
  role emotional 3 months | 78.0 (37.6) | 74.5 (38.4)
  role emotional 6 months | 89.4 (26.7) | 82.8 (34.5)
  role emotional 12 months | 90.7 (25.8) | 89.3 (25.3)
  role emotional 24 months | 92.2 (20.9) | 88.2 (27.5)
  Mental health baseline | 79.0 (13.9) | 78.5 (13.4)
  Mental health 6 weeks | 79.5 (15.6) | 76.3 (15.4)
  Mental health 3 months | 79.8 (15.8) | 82.4 (12.8)
  Mental health 6 months | 81.9 (13.8) | 83.9 (12.4)
  Mental health 12 months | 82.8 (15.0) | 83.1 (12.2)
  Mental health 24 months | 81.4 (14.8) | 84.1 (12.0)

5. Secondary Outcome: Adverse Events
Description: The following complications were monitored throughout study:
  * Medical related: urinary, gastrointestinal, cardiac, pulmonary, metabolic
  * Surgical related: nerve injury, superficial or deep infection, dislocation, frozen shoulder, hematoma, biceps rupture, failure of tendon healing, dermatitis, reflex sympathetic dystrophy (RSD), persistent pain, re-injury.
  * Other
  The surgeon responsible for the patient used clinical judgment to make a decision regarding if the complication was related or not to the treatment being tested (use or not of sling).
Time Frame: 2 weeks, 6 weeks, 3 months, 6months
Population: Expected, surgical procedure related: superficial infection, frozen shoulder, biceps rupture, persistent pain, reinjury Unexpected, not treatment related: Traumatic reinjury
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Early ROM) | Group B (Usual Care)
Number analyzed (Participants) | 87 | 89
Participants
  Superficial Infection | 0 | 1
  Frozen Shoulder | 1 | 2
  Biceps Rupture | 1 | 1
  Persistent Pain | 10 | 6
  Re-injury not requiring surgery | 5 | 4
  Urinary | 0 | 0
  Gastrointestinal | 0 | 0
  Cardiac | 0 | 0
  Pulmonary | 0 | 0
  Metabolic | 0 | 0
  Nerve Injury | 0 | 0
  Deep infection | 0 | 0
  Dislocation | 0 | 0
  Hematoma | 0 | 0
  Dermatitis | 0 | 0
  Reflex Sympathetic Dystrophy (RSD) | 0 | 0
  Traumatic Re-injury | 0 | 2

6. Secondary Outcome: Pain in the Shoulder at Baseline, 6 Weeks, 3, 6, 12, 24 Months
Description: Shoulder pain at rest, with activity and at night were measured using a visual analogue scale of 0-10 (no pain to severe pain)
Time Frame: baseline, 6 weeks, 3, 6, 12, 24 months
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Group A (Early ROM) | Group B (Usual Care)
Number analyzed (Participants) | 87 | 89
centimeters
  Pain at rest - baseline | 3.1 (2.3) | 2.9 (2.4)
  Pain at rest 6 weeks | 2.2 (2.0) | 2.0 (1.9)
  Pain at rest 3 months | 1.8 (2.1) | 1.4 (1.6)
  Pain at rest 6 months | 0.9 (1.3) | 0.8 (1.0)
  Pain at rest 12 months | 0.6 (1.0) | 0.6 (1.0)
  Pain at rest 24 months | 0.7 (1.3) | 0.6 (1.3)
  Pain with activity - baseline | 6.1 (2.4) | 5.8 (2.3)
  Pain with activity 6 weeks | 4.4 (2.5) | 3.9 (2.1)
  Pain with activity 3 months | 3.4 (2.4) | 2.8 (1.9)
  Pain with activity 6 months | 2.2 (1.9) | 1.8 (1.5)
  Pain with activity 12 months | 1.2 (1.4) | 1.2 (1.4)
  Pain with activity 24 months | 1.2 (1.6) | 1.0 (1.6)
  Pain at night - baseline | 4.8 (2.6) | 4.4 (2.7)
  Pain at night 6 weeks | 3.3 (2.5) | 2.8 (2.1)
  Pain at night 3 months | 2.3 (2.4) | 2.1 (2.0)
  Pain at night 6 months | 1.1 (1.6) | 1.0 (1.2)
  Pain at night 12 months | 0.6 (0.8) | 0.8 (1.4)
  Pain at night 24 months | 0.9 (1.6) | 0.7 (1.4)

ADVERSE EVENTS:
Time Frame: Over 24 months
Arm/Group | Group A (Early ROM) | Group B (Usual Care)
All-Cause Mortality (participants affected / at risk) | 0/103 | 0/103
Serious Adverse Events (participants affected / at risk) | 0/103 | 0/103
Other Adverse Events (participants affected / at risk) | 10/103 | 6/103
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (Early ROM) (N=103) | Group B (Usual Care) (N=103)
Persistent Pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 6 (6) — Pain in the surgical shoulder that needed further intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No